CLINICAL TRIAL: NCT04138797
Title: Evaluation of Non-invasive Measurement of Electrophysiological "HV" Interval Using a High-density and High-fidelity Signal Averaging ECG Device
Acronym: BIOSEMI-HV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2019/11
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Cardiac Electrophysiology; Electrocardiogram
Keywords: Signal Averaging ECG; HV interval

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electrophysiological exploration & ECG Biosemi (Experimental)
  Interventions: Procedure: Electrophysiological exploration; Device: ECG Biosemi

INTERVENTIONS:
Procedure: Electrophysiological exploration — Electrophysiological exploration is performed, as part of the routine care, after the Biosemi high density ECG, the same day or maximum 4 days later. It is performed in interventional rhythmology room, under fluoroscopic control. After local anesthesia, one or more introducers are placed in the femoral vein allowing the introduction of catheters. These catheters allow recording of the HV interval
Device: ECG Biosemi — Non invasive ECG monitoring for HV measurement using high density Biosemi device. This device use 256 skin electrodes. At the same time and with the same system, a chest pressure sensor can record the patient's breathing movements.

SUMMARY:
His-Ventricle (HV) measurement is only obtained invasively using transvenous catheters. This kind of procedure is routinely performed but some risks of complication exist. HV interval prolongation is correlated with increased risk of occurrence of complete atrioventricular block which could lead to syncope or cardiac sudden death. A new non invasive, high density and high fidelity system (BioSemi, BioSemi B.V., Amsterdam, Netherlands) can theorically collect such electrophysiological signal using a signal averaging acquisition method. We want to assess the possibility of non invasive HV interval measurement using this new device.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted at Bordeaux University Hospital for electrophysiological study with HV measurement.

Exclusion Criteria:

* Patients under 18 years old,
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Measurement of HV interval correlation by the intra-class correlation coefficient | Day 0
  The correlation of the HV interval obtained using the 2 different methods, is measured by a correlation coefficient
Measurement of HV interval correlation by graphical representation | Day 0
  The correlation of the HV interval obtained using the 2 different methods, is measured by a graphical representation of Bland and Altman

CONTACTS AND LOCATIONS:
Overall Officials: Josselin DUCHATEAU, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Pessac, France